CLINICAL TRIAL: NCT06793098
Title: Assessment of the Concentrations of Functional Proteins as Potential Early Markers of Insulin Resistance in Women With Polycystic Ovary Syndrome
Brief Title: Functional Proteins in Polycystic Ovary Syndrome
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, PhD, MD, Principal Investigator, Jagiellonian University
Other Study IDs: 1072.6120.44.2024-3
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Reproductive Age; PCOS (Polycystic Ovary Syndrome)
Keywords: insulin resistance; kisspeptin; ghrelin; zonulin; metabolic syndrome; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women with polycystic ovary syndrome (PCOS) and insulin resistance (IR)
  Interventions: Diagnostic Test: Measurement of kisspeptin concentration; Diagnostic Test: Measurement of ghrelin concentration; Diagnostic Test: Measurement of zonulin concentration
- Women with polycystic ovary syndrome (PCOS) without insulin resistance (IR)
  Interventions: Diagnostic Test: Measurement of kisspeptin concentration; Diagnostic Test: Measurement of ghrelin concentration; Diagnostic Test: Measurement of zonulin concentration
- Women without PCOS
  Interventions: Diagnostic Test: Measurement of kisspeptin concentration; Diagnostic Test: Measurement of ghrelin concentration; Diagnostic Test: Measurement of zonulin concentration

INTERVENTIONS:
Diagnostic Test: Measurement of kisspeptin concentration — Measurement of kisspeptin concentration in fasting venous blood serum
Diagnostic Test: Measurement of ghrelin concentration — Measurement of ghrelin concentration in fasting venous blood serum
Diagnostic Test: Measurement of zonulin concentration — Measurement of zonulin concentration in fasting venous blood serum

SUMMARY:
The concentration of functional proteins: kisspeptin, ghrelin, zonulin will be measured and compared in women with polycystic ovary syndrome (PCOS) and insulin resistance (IR), in women with PCOS without IR, and in women without PCOS.

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS) is currently the most common endocrine disorder in women of reproductive age with an unknown etiology. A predominant metabolic feature of PCOS is insulin resistance (IR), which contributes to the pathogenesis and expression of other symptoms of the syndrome, such as hyperandrogenism. The metabolic disturbances in women with PCOS result in a higher incidence of cardiovascular diseases and endometrial cancer in the premenopausal age. The gold standard for assessing peripheral tissue sensitivity to insulin is the hyperinsulinemic-euglycemic clamp technique; however, this method is not commonly used in clinical practice due to its complexities. Instead, simpler tests, such as the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) and fasting insulin measurements along with glucose tolerance tests, are employed. These methods are utilized for diagnosing insulin resistance rather than identifying predispositions. Therefore, there is an urgent need to identify more precise markers of IR that could be used in routine early-stage assessments. Given the long-term complications associated with PCOS, which can shorten life expectancy, early diagnosis and treatment of IR are crucial. Furthermore, such studies may contribute to exploring the etiopathogenesis of the syndrome. The discovery of "markers" that can predict or diagnose metabolic abnormalities at an early stage, prior to the onset of clinical symptoms, would facilitate early intervention and treatment, thus preventing a decline in quality of life associated with PCOS.

This study will measure and compare the concentrations of locally acting hormones: ghrelin, kisspeptin, and zonulin in three research groups: women with polycystic ovary syndrome (PCOS) and insulin resistance (IR), women with PCOS without IR, and women without PCOS. Measurements will be performed using immunoenzymatic methods (ELISA) and the Erba XL biochemical analyzer. Statistical calculations will be conducted using SPSS Statistics software.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-45 years

Exclusion Criteria:

* removal of at least one ovary
* treated diabetes of any type
* diagnosed and treated metabolic diseases
* diagnosed and treated autoimmune diseases
* diagnosed and treated autoinflammatory diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women aged 18-45 years managed for menstrual irregularities or for routine check-up
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement and comparison of kisspeptin concentrations expressed in [pg/ml] in all three study groups | up to 6 months
Measurement and comparison of ghrelin concentrations expressed in [pg/ml] in all three study groups | up to 6 months
Measurement and comparison of zonulin concentrations expressed in [pg/ml] in all three study groups | up to 6 moths

CONTACTS AND LOCATIONS:
Overall Officials: Kazimierz Pityński, Prof., Ph.D., M.D., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University, Krakow, Poland